CLINICAL TRIAL: NCT03630016
Title: SpO2 Accuracy Comparison of Smart Sock V. 2 SpO2 to Arterial Blood CO-Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Owlet Baby Care, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR2017-263
Record Dates: First submitted 2018-08-03; First posted 2018-08-14 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia | interventions — Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Reference CO-Oximetry (Active Comparator): Reference Co-Oximetry
  Interventions: Diagnostic Test: Pulse oximetry with Owlet BabySat v1.0 sensor
- Owlet BabySat v1.0 (Experimental): Owlet BabySat v1.0
  Interventions: Diagnostic Test: Pulse oximetry with Owlet BabySat v1.0 sensor
- Owlet Smart Sock V2 v1.1 (Experimental): Owlet Smart SockTM 2 , OSS v1.1 Sensor and Custom Adult Thumb Sock
  Interventions: Diagnostic Test: Pulse oximetry with Owlet BabySat v1.0 sensor

INTERVENTIONS:
Diagnostic Test: Pulse oximetry with Owlet BabySat v1.0 sensor — A comparative, single-center, non-randomized study to evaluate the SpO2 accuracy guidelines for pulse oximetry over the range of 70-100% SaO2 under non-motion conditions. Arterial blood sampling measured by functional SaO2 CO-Oximetry, was used as the basis for comparison with Owlet BabySat v1.0 and Owlet Smart Sock 2 sensors

SUMMARY:
Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians in everyday situations to estimate arterial oxygen saturation. There are two devices used in this investigational study: BabySat v.1.0 and Owlet Baby Care, Inc. Smart SockTM 2 (currently available over-the-counter), with specific emphasis on its pulse oximetry accuracy. The BabySat and Smart SockTM 2 are non-invasive home care devices for use with infants. The purpose of this study was to validate the SpO2 accuracy of BabySat v1.0 and Owlet Smart SockTM 2, OSS v1.1 sensors pulse oximetry, during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry.

DETAILED DESCRIPTION:
Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians in everyday situations to estimate arterial oxygen saturation. A pulse oximeter is a device that measures the oxygen saturation of arterial blood non-invasively.

The purpose of this study was to evaluate the SpO2 accuracy performance of the Owlet BabySat v1.0 and Smart SockTM 2 pulse oximetry OSS v1.1 sensors during non-motion conditions over the range of 70-100% SaO2 to arterial blood samples assessed by CO-Oximetry for a SpO2 validation.

The goal, in its entirety, was to show the SpO2 accuracy performance for the investigational device Owlet Baby Care, Inc. Smart SockTM V. 2.

It was expected that the Accuracy Root Mean Square (ARMS) performance would meet the required specification of ARMS 3% or lower in non-motion conditions for the range of 70 - 100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification.

No risks or adverse device effects were expected. There were no contraindications for use in the proposed study population.

The study was conducted in accordance to the code of federal regulations for non-significant risk medical device studies and applicable ISO 14155 (2nd edition 2011-02-01), applicable sections of ISO80601-2-61 (1st edition 2011-04- 01), and Pulse Oximeters - Premarket Notifications Submissions [510(k)s] Guidance For Industry and Food and Drug Administration Staff (issued: March 4, 2013)

ELIGIBILITY:
Inclusion Criteria:

* 10-15 Adults with a minimum of 3 males and a minimum of 3 females, with the balance, made up of either.
* Subject must have the ability to understand and provide written informed consent
* Subject is 18 to 50 years of age
* At least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who have not smoked within 2 days prior to the study.

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study
* Females who are pregnant, who are trying to get pregnant
* Smoker Subjects who have refrained will be screened for COHb levels
* Subjects with known heart or cardiovascular conditions
* Subjects with known clotting disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milena Adamian, MD, Study Director — Owlet Baby Care, Inc.
Locations (1):
- Owlet Baby Care, Inc., Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eleven subjects were enrolled into the study with one subject later withdrawn due to poor sensor placement.
Period: Overall Study
Arm/Group | Owlet Smart Sock V2 v1.1
Started | 11
Completed | 10
Not Completed | 1
Not completed — Poor Sensor Placement | 1

BASELINE CHARACTERISTICS:
Arm/Group | Owlet Smart Sock V2 v1.1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Weight [Mean (Standard Deviation); unit: lbs] | 159.8 (25.8)
Height [Mean (Standard Deviation); unit: inches] | 68.1 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: It Was Expected That the Accuracy Root Mean Square (ARMS) Between Measured SpO2 of Owlet Smart Sock V2 v1.1 and Reference SpO2 Would Meet the Required Specification of ARMS 3% or Lower in Non-motion Conditions for the Range of 70 - 100%
Description: The purpose of the study was to evaluate the accuracy of the blood oxygen saturation (SpO2) at rest over the range of 70-100% compared to arterial blood samples assessed by standard methods [Co-Oximetry]. A standard pulse oximeter accuracy is evaluated by the Accuracy Root Mean Square (ARMS). The results of accurate performance of the oximetry system require ARMS of 3% or less in non-motion conditions for the range of 70-100% SpO2 per standard.
Time Frame: Acute immediate assessment of the sensor accuracy compared to CO-oximetry
Measure: Number; unit: Percent SpO2
Units Other Than Participants: Number of Data Points
Arm/Group | Owlet Smart Sock V2 v1.1
Number analyzed (Participants) | 10
Number analyzed (Number of Data Points) | 226
Percent SpO2 | 2.4

ADVERSE EVENTS:
Time Frame: Throughout study duration and a follow-up with each subject will be conducted within 7 days following participation in the study and will be conducted via telephone, text or email.
Arm/Group | Owlet Smart Sock V2 v1.1
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT03630016/Prot_SAP_000.pdf